CLINICAL TRIAL: NCT00584415
Title: Navi-Star Thermo-Cool Catheter For Ablation of Atrial Fibrillation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 010971
Record Dates: First submitted 2007-12-20; First posted 2008-01-02 (Estimated); Results first posted 2014-07-28 (Estimated); Last update posted 2014-07-28 (Estimated); Status verified 2014-07

CONDITIONS: Paroxysmal Atrial Fibrillation
Keywords: Catheter Ablation; Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- GP + PVI ablation (Active Comparator): This study contains only one arm, which is GP ablation + PV antrum isolation. The intervention (GP ablation + PV isolation) was performed using ThermoCool Navistar catheters in all patients
  Interventions: Device: GP ablation + PV isolation

INTERVENTIONS:
Device: GP ablation + PV isolation — All patients underwent GP ablation and PV isolation using the NaviStar ThermoCool ablation catheter
  Other Names: Navi-Star ThermoCool Catheter, Biosense-Webster Inc.

SUMMARY:
The objective of this study is to demonstrate that the NAVI-STAR THERMO-COOL catheter can be used to safely and effectively reduce symptomatic episodes of paroxysmal atrial fibrillation in patients with frequent (>3 episodes/month) or infrequent <3 episodes/month)atrial fibrillation resistant to at least one Class I or Class III antiarrhythmic drug.

DETAILED DESCRIPTION:
The ability of a saline irrigated catheter to deliver RF energy at higher power with a lower electrode-tissue interface temperature, combined with the anatomical guidance of electroanatomical mapping should allow:

1. Isolation of the pulmonary veins at the LA-PV junction with the same or lower risk of pulmonary vein stenosis;
2. Creation of continuous, transmural linear left atrial lesions with the same or lower risk of thromboembolism;
3. These two factors will eliminate documented episodes of symptomatic sustained AF in patients with frequent (>3 episodes/month) or infrequent (<3 episodes/month);
4. Patients with interruption of the vagal response (sinus bradycardia or AV block) during stimulation at the sites of left atrial autonomic ganglionated plexi (GP) will have lower recurrence of atrial fibrillation.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater or equal to 18 years
2. At least one documented episode of atrial fibrillation (AF) within the previous 6 months.
3. Failure of at least one antiarrhythmic drug (Class I or III) defined as recurrence of AF or adverse effect.
4. Informed consent obtained.

Exclusion Criteria:

1. Left atrial thrombus
2. Acute myocardial infarction within eight (8) weeks
3. Atriotomy within eight (8) weeks
4. Decompensated heart failure (unless the AF is thought to be a significant etiologic factor and AF ablation is clinically indicated)
5. Pregnancy
6. Ablation in a pulmonary vein within 4 months.
7. Occurrence of perforation during an ablation procedure performed less than two months prior to the planned ablation date.
8. Significant congenital anomaly or medical problem that, in the opinion of the investigator, would preclude enrollment in the study.
9. Enrolled in an investigational study evaluating another device or drug
10. Unwilling to participate in the study or unavailable for follow-up visits.
11. Incarcerated

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2004-02; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sunny Po, MD, Principal Investigator — University of Oklahoma
Locations (1):
- University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- GP Ablation + PV Isolation: All patients in this study received pulmonary vein isolation (PVI) and ganglionated plexi (GP) ablation to treat paroxysmal AF
Period: Overall Study
Arm/Group | GP Ablation + PV Isolation
Started | 119 (A total of 119 enrolled and 112 underwent the ablation procedure;)
Completed | 112
Not Completed | 7
Not completed — Adverse Event | 7

BASELINE CHARACTERISTICS:
Groups:
- PV Isolation + GP Ablation: All patients received pulmonary vein antrum isolation (PV isolation) and ablation of the major atrial ganglionated plexi (superior left GP, inferior left GP, anterior right GP and inferior right GP). Ganglionated plexi (GP) were identified by delivering high-frequency stimulation (20 Hz) from the ablation catheter. If vagal response (AV block) was initiated by stimulation, that site was counted as a GP site and was then ablated.
Arm/Group | PV Isolation + GP Ablation
Number analyzed (Participants) | 119
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 95
  >=65 years | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 92
Region of Enrollment [Number; unit: participants]
  United States | 119

OUTCOME MEASURES:

1. Primary Outcome: Atrial Tachyarrhythmia Recurrence in Participants
Description: Outcome is determined by recurrence of atrial tachyarrhythmia in participants. Outcome is measured by any atrial tachyarrhythmias recorded by 12-lead ECGs, Holter monitoring or event monitoring. Recurrence of atrial tachyarrhythmia is also measured by symptoms reported by patients. Symptoms include palpitations, dizziness, dyspnea and any AF-related symptoms that existed before AF ablation.
Time Frame: 0-5 years
Population: all patients referred for paroxysmal AF ablation between 1-2004 and 12-2005 were included
Measure: Number; unit: participants
Groups:
- GP Ablation + PV Isolation): All patients received high-frequency stimulation (20 Hz) to the presumed GP site to elicit a vagal response (AV block). After all GP sites were ablated, all patients underwent circumferential PV isolation.
Arm/Group | GP Ablation + PV Isolation)
Number analyzed (Participants) | 119
participants | 37

2. Secondary Outcome: Total Number of Significant Ablation Procedure Related Complications
Description: Any complication directly related to the ablation procedure was included. These complications included pericardial effusion, cardiac tamponade, excessive bleeding requiring transfusion, phrenic nerve injury, atrio-esophageal fistula, vascular access complications, myocardial infarction and stroke.
Time Frame: 0-1 year
Measure: Number; unit: Complications
Groups:
- Experimental Arm (GP Ablation + PV Antrum Isolation): All patients received high-frequency stimulation (20 Hz) to the presumed GP site to elicit a vagal response (AV block). After all GP sites were ablated, all patients underwent circumferential PV isolation.
Arm/Group | Experimental Arm (GP Ablation + PV Antrum Isolation)
Number analyzed (Participants) | 119
Complications | 10

ADVERSE EVENTS:
Time Frame: The adverse effects were collected within the 1st year after ablation.
Arm/Group | Experimental Arm (GP Ablation + PV Antrum Isolation)
Serious Adverse Events (participants affected / at risk) | 10/119
Other Adverse Events (participants affected / at risk) | 9/119
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental Arm (GP Ablation + PV Antrum Isolation) (N=119)
serious (Cardiac disorders) | 10 (10)
pericardial effusion/tamponade (Cardiac disorders) | 7 (7)
stroke (Nervous system disorders) | 1 (1)
phrenic nerve injury (Nervous system disorders) | 1 (1)
death (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental Arm (GP Ablation + PV Antrum Isolation) (N=119)
groin hematoma (Vascular disorders) | 6 (6)
pneumonia (Infections and infestations) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes